CLINICAL TRIAL: NCT02015884
Title: Impact of a Program to Prevent the Risk of Antisocial Behavior and Attacks of Patients or Attendant on Healthcare Workers in an Ophthalmic Emergency Unit.
Brief Title: Antisocial Behavior on Healthcare Professionals in an Emergency Unit.
Acronym: PREVURGO
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: D50794
Record Dates: First submitted 2013-12-10; First posted 2013-12-19 (Estimated); Last update posted 2015-10-23 (Estimated); Status verified 2015-10

CONDITIONS: Rudeness/Incivility, Aggression or Violence Against Healthcare Workers in an Ophthalmic Emergencies Unit.
Keywords: Incivility; Rudeness; Aggression; Violent act; Healthcare workers; Emergency unit
MeSH Terms: conditions — Incivility; Aggression; Emergencies

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All patients admitted to the ophthalmologic emergency unit.

SUMMARY:
At the hospital, the attacks against health professionals are becoming commonplace, making working conditions difficult. The ophthalmological emergencies are a perfect testing ground to evaluate the effectiveness of a series of original actions to prevent the occurrence of violence against healthcare workers. The main objective is to measure the impact of an integrated prevention of the occurrence of antisocial behavior or attacks against the healthcare workers.

The prevention program combines five interventions (steps): 1) a computer sorting algorithm and specific screens for calling patients in waiting rooms, 2) a clear signage to direct patients between waiting rooms, treatment rooms and administrative et medical offices, 3) Posts information on the activity of emergency services displayed on screens, in the waiting rooms, 4) a mediator/go-between/conciliator, 5) and a dummy surveillance camera.

This is an interrupted time series study. All patients admitted to the ophthalmological emergency unit of a university hospital located in Lyon, France, are included in the study, from June 2013 to Sept 2015

ELIGIBILITY:
Inclusion Criteria:

* Patient admitted to the ophthalmologic emergency unit

No Exclusion Criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients admitted to the ophthalmologic emergency unit will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 58465 (Actual)
Dates: Start 2013-05; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Proportion of patients (or their attendants) who committed a rudeness/incivility or aggression or violence against healthcare workers. | Patients will be followed for the duration of the ophthalmic emergency unit stay, an expected average of 2 hours.
  When seeking to characterize the violent behavior, three levels of increasing aggressiveness are typically distinguished: a) incivility i.e. the lack of respect for others characterized by relatively mild acts, b) physical or verbal aggression (insults, threats, assault), and c) the violent act.

SECONDARY OUTCOMES:
Occurrence of antisocial behavior or assaults against other patients or carers attending the ophthalmological emergencies. | Patients will be followed for the duration of the ophthalmic emergency unit stay, an expected average of 2 hours.
  Proportion of incivility or assaults against other patients or attendant present (number of incivility or assaults on the number of patients admitted to the emergency)
Waiting times for patients | Patients will be followed for the duration of the ophthalmic emergency unit stay, an expected average of 2 hours.
  Average waiting times for patients with ophthalmic emergencies before they were taken care of by a doctor.
Stress of healthcare personnel | 30 minutes
  Stress at work of health personnel engaged in an ophthalmic emergency unit measured by the Karasek questionnaire. 30 mn are necessary to complete the questionnaire.
Satisfaction of patients | Patients will be followed for the duration of the ophthalmic emergency unit stay, an expected average of 2 hours.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon - Hôpital Edouard Herriot, Lyon, France

REFERENCES:
- [Derived] Touzet S, Occelli P, Denis A, Cornut PL, Fassier JB, Le Pogam MA, Duclos A, Burillon C. Impact of a comprehensive prevention programme aimed at reducing incivility and verbal violence against healthcare workers in a French ophthalmic emergency department: an interrupted time-series study. BMJ Open. 2019 Sep 5;9(9):e031054. doi: 10.1136/bmjopen-2019-031054. PMID 31492791
- [Derived] Touzet S, Cornut PL, Fassier JB, Le Pogam MA, Burillon C, Duclos A. Impact of a program to prevent incivility towards and assault of healthcare staff in an ophtalmological emergency unit: study protocol for the PREVURGO On/Off trial. BMC Health Serv Res. 2014 May 19;14:221. doi: 10.1186/1472-6963-14-221. PMID 24885544